CLINICAL TRIAL: NCT04414007
Title: The Application of Internet+ Home-based Cardiac Rehabilitation Model in Atrial Fibrillation Patients After Radio Frequency Ablation
Brief Title: The Application of Internet+ Home-based Cardiac Rehabilitation in Atrial Fibrillation Patients After RFCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Zhipeng BAO, Principal Investigator, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2020-SR-038
Record Dates: First submitted 2020-05-27; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Atrial Fibrillation; Cardiac Rehabilitation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet+ home-based cardiac rehabilitation group (Experimental): The Internet+ home-based cardiac rehabilitation group receive home-based cardiac rehabilitation program through Internet platform and intelligent wearable devices .
  Interventions: Behavioral: Internet+ home-based cardiac rehabilitation
- conventional care group (Active Comparator): The UC-assigned patients will maintain standard of care.The conventional rehabilitation group received routine medical care and traditional home-based cardiac rehabilitation based on the rehabilitation manual and exercise diary, followed up by telephone and outpatient.
  Interventions: Behavioral: Conventional rehabilitation

INTERVENTIONS:
Behavioral: Internet+ home-based cardiac rehabilitation — The Internet+ home-based cardiac rehabilitation group receive home-based cardiac rehabilitation program through Internet platform and intelligent wearable devices .
  Arms: Internet+ home-based cardiac rehabilitation group
Behavioral: Conventional rehabilitation — We provide patients with cardiac rehabilitation manuals and exercise logs. 4 weeks after ablation，Patients have CPET.Their exercise prescription was made according to CPET .The patients have rehabilitation training at home and recorded their exercise data including exercise time、type、frequency and average heart rate.
  Arms: conventional care group

SUMMARY:
Epidemiological reports show that the incidence of atrial fibrillation continues to increase. AF is the most common arrhythmia with high mortality and disability rate. Radio frequency ablation has good therapeutic effect of AF symptoms. However, even after successful radio frequency ablation, there are still many discomforts that deserve medical attention. The benefits of cardiac rehabilitation for patients with heart disease have been recognized，but the adherence with cardiac rehabilitation is not satisfactory. Home-based rehabilitation has received increasing recognition because it has overcome many obstacles for patients to participate in cardiac rehabilitation. The application of Internet+ follow-up mode and intelligent wearable devices provide new ideas for home-based cardiac rehabilitation with the progress of information technology nowadays. This study used an experimental research design. The aim was to explore the application effects of Internet platform and wearable devices in home-based cardiac rehabilitation in patients with atrial fibrillation after radio frequency ablation. The final goal is to provide the basis for the development and application of this kind of home-based cardiac rehabilitation care in patients with atrial fibrillation after radio frequency ablation.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with atrial fibrillation and planned for treatment with radiofrequency catheter ablation (RFA) for AF;
* Patients with age from 18 to 75 years;
* Patients or primary caregiver are able to use smartphones;
* Providing oral and written informed consent.

Exclusion Criteria:

* Radiofrequency ablation was not performed for various reasons;
* patients who were unable to understand the study due to severe cognitive impairment;
* Patients with psychiatric disorders;
* Patients with serious and instable body or severe complications;
* Patients sufferring other exercise contraincations.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
6-minute walk test | Change from Baseline 6-minute walk distance at 2 years
  exercise capacity
Peak VO2 | Change from Baseline Peak VO2 at 2 years
  exercise capacity
sf-36 | Change from Baseline sf-36 at 2 years
  Quality of Life

SECONDARY OUTCOMES:
SAS | Change from Baseline SAS scores at 2 years
  Anxious
SDS | Change from Baseline SDS scores at 2 years
  Depression
PSQI | Change from Baseline PSQI scores at 2 years
  sleep quality
EHRA score | Change from Baseline EHRA scores at 2 years
  AF burden
AF recurrence | Change from Baseline AF recurrence at 2 years
  patients still have episode of atrial fibrillation three months after ablation
Adherence | at 2 years
  Percentage of completed exercise prescription weeks

CONTACTS AND LOCATIONS:
Overall Officials: Guozhen Sun, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated hospital of Nanjing Medical University, Najing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No